CLINICAL TRIAL: NCT04894136
Title: Reproductive and Obstetric Outcomes in TESE-ICSI Cycles: a Comparison Between Obstructive and Non-obstructive Azoospermia
Brief Title: Reproductive and Obstetric Outcomes in TESE-ICSI Cycles for Azoospermia
Acronym: AZOOCOMES
Status: Completed | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: 1906
Record Dates: First submitted 2021-04-16; First posted 2021-05-20 (Actual); Last update posted 2021-05-20 (Actual); Status verified 2021-03

CONDITIONS: Obstructive Azoospermia; Non-obstructive Azoospermia; Obstetric Complication
Keywords: Reproductive outcomes
MeSH Terms: interventions — Embryo Transfer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ICSI-TESE cycles for obstructive azoospermia: Couples who underwent ICSI-TESE cycles for obstructive azoospermia between January 2001 and December 2019 at Humanitas Fertility Center
  Interventions: Procedure: ICSI-TESE; embryo-transfer
- ICSI-TESE cycles for nonobstructive azoospermia: Couples who underwent ICSI-TESE cycles for nonobstructive azoospermia between January 2001 and December 2019 at Humanitas Fertility Center
  Interventions: Procedure: ICSI-TESE; embryo-transfer

INTERVENTIONS:
Procedure: ICSI-TESE; embryo-transfer — The sperm injected into the cytoplasm of an oocyte (Intracytoplasmatic Sperm Injection) is obtained by testicular extraction. Ultrasound guided transvaginal embryo transfer.

SUMMARY:
A comparison of reproductive and obstetrical outcomes is retrospectively performed among couples that underwent ICSI-TESE cycles for obstructive and non obstructive azoospermia between January 2001 and December 2019.

DETAILED DESCRIPTION:
Azoospermia affects almost 20% of all infertile males and It can be divided into obstructive azoospermia (OA) and nonobstructive azoospermia (NOA). Assisted fertilization with testicular sperm extraction (TESE) and intracytoplasmatic sperm injection (ICSI) has been successfully applied for its treatment.

Review of the literature shows that there is a lack of consensus about reproductive outcomes between men with OA and NOA. No study has ever investigated differences in obstetrical outcomes between these two groups before.

The objective of this study is to retrospectively determine differences in reproductive and obstetrical outcomes among couples that underwent ICSI-TESE cycles for obstructive and non obstructive azoospermia.

The primary outcomes that will be investigated include:

* Reproductive outcomes: pregnancy rate, live birth rate (LBR) and abortion rate.
* Obstetrical outcomes: twinning rate, gestational age, prematurity rate, birth weight, cesarean section rate and the rate of the main obstetrical complication, such as pre-eclampsia, gestational hypertension, intrauterine growth restriction (IUGR).

ELIGIBILITY:
Inclusion Criteria for obstructive azoospermia group:

* infertility
* diagnosis of obstructive azoospermia
* ICSI-TESE cycles

Inclusion Criteria for non-obstructive azoospermia group:

* infertility
* diagnosis of non-obstructive azoospermia
* ICSI-TESE cycles

Exclusion Criteria:

* Sperm donation
* Use of ejaculated sperm
* Couples who underwent pre-implantation genetic testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study database will include all the couples who underwent ICSI-TESE cycles between January 2001 and December 2019 at Humanitas Fertility Center after ICSI-TESE for obstructive and nonobstructive azoospermia.
  ICSI-TESE cycles not reaching the stage of oocyte retrieval will be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 520 (Actual)
Dates: Start 2001-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Live birth rate (LBR) | 20 years (2001-2019)
  Rate of delivery of a living baby after at least 22 weeks of gestation
Pregnancy rate | 20 years (2001-2019)
  Total number of pregnancies including live births, abortions and fetal death
Abortion rate | 20 years (2001-2019)
  Proportion of clinical pregnancies who failed to continue beyond 22 weeks of gestation
Maternal complications rate | 20 years (2001-2019)
  Incidence of the obstetric complications, such as pre-eclampsia, gestational hypertension, placenta previa and placental abruption, intrauterine growth restriction.
Gestational age | 20 years (2001-2019)
  Mean gestational age of the pregnancies considered (written with both weeks and days)
Prematurity rate | 20 years (2001-2019)
  Rate of pregnancies lasted less than 37 weeks and 0 days
Twinning rate | 20 years (2001-2019)
  Rate of twin deliveries out of the total number of deliveries
Cesarean section rate | 20 years (2001-2019)
  Rate of cesarean section deliveries out of the total number of deliveries
Birth weight | 20 years (2001-2019)
  Mean birth weight of the neonates written in grams.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bocca S, Moussavi V, Brugh V, Morshedi M, Stadtmauer L, Oehninger S. ICSI outcomes in men undergoing TESE for azoospermia and impact of maternal age. Andrologia. 2017 Mar;49(2). doi: 10.1111/and.12617. Epub 2016 May 20. PMID 27198124
- [Background] He X, Cao Y, Zhang Z, Zhao J, Wei Z, Zhou P, Cong L. Spermatogenesis affects the outcome of ICSI for azoospermic patients rather than sperm retrieval method. Syst Biol Reprod Med. 2010 Dec;56(6):457-64. doi: 10.3109/19396368.2010.513078. Epub 2010 Oct 14. PMID 20942727
- [Background] La Sala GB, Valli B, Leoni S, Pescarini M, Martino F, Nicoli A. Testicular sperm aspiration (TESA) in 327 ICSI cycles. Int J Fertil Womens Med. 2006 Jul-Aug;51(4):177-82. PMID 17184103
- [Background] Palermo GD, Schlegel PN, Hariprashad JJ, Ergun B, Mielnik A, Zaninovic N, Veeck LL, Rosenwaks Z. Fertilization and pregnancy outcome with intracytoplasmic sperm injection for azoospermic men. Hum Reprod. 1999 Mar;14(3):741-8. doi: 10.1093/humrep/14.3.741. PMID 10221707